CLINICAL TRIAL: NCT00674817
Title: A Randomized, Double-blind, Crossover Study to Investigate the Bronchodilatation Post-inhalation of GSK961081 Alone and With the Addition of Cumulative Doses of Short Acting Bronchodilators (Salbutamol and Ipratropium Bromide) in Patients With COPD
Brief Title: An Investigation Of The Interaction Of GSK961081 With Inhaled Beta-Agonist And Anti-Muscarinic Drugs.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MAB110123
Record Dates: First submitted 2008-04-24; First posted 2008-05-08 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: salbutamol,; Chronic Obstructive Pulmonary Disease (COPD); GSK961081 muscarinic receptor antagonist,; COPD; ipratropium bromide,; Asthma; ß2-adrenergic agonist,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 400 microgrammes GSK961081 and salbutamol (Experimental): 400 microgrammes of GSK961081 single-dose (via DISKUS Metered Dry Powder Inhaler/ MDPI) followed by cumulative doses (3x 200 microgrammes at 20 min intervals, administered via spacer) of salbutamol at 1h, 12h and 24h of dosing.
  Interventions: Drug: 400 microgrammes GSK961081
- 1200 microgrammes GSK961081 and salbutamol (Experimental): 1200 microgrammes of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (3x 200 microgrammes at 20 min intervals, administered via spacer) of salbutamol at 1h, 12h and 24h of dosing.
  Interventions: Drug: 400 microgrammes GSK961081; Drug: 1200 microgrammes GSK961081
- 400 microgrammes GSK961081 and ipratropium bromide (Experimental): 400 microgrammes of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (20 microgrammes, 20 microgrammes and 40 microgrammes at 20 min intervals, administered via spacer) of ipratropium bromide at 1h, 12h and 24h of dosing.
  Interventions: Drug: 1200 microgrammes GSK961081
- 1200 microgrammes of GSK961081 and ipratropium bromide (Experimental): 1200 microgrammes of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (20 microgrammes, 20 microgrammes and 40 microgrammes at 20 min intervals, administered via spacer) of ipratropium bromide at 1h, 12h and 24h of dosing.
  Interventions: Drug: 400 microgrammes GSK961081; Drug: 1200 microgrammes GSK961081
- 400 microgrammes of GSK961081 and placebo (Placebo Comparator): 400 microgrammes of GSK961081 single-dose (via DISKUS Metered Dry Powder Inhaler/ MDPI) followed by cumulative doses (3 doses at 20 min intervals, administered via spacer) of placebo at 1h, 12h and 24h of dosing.
  Interventions: Drug: 1200 microgrammes GSK961081
- 1200 microgrammes of GSK961081 and placebo (Placebo Comparator): 1200 microgrammes of GSK961081 single-dose (via DISKUS Metered Dry Powder Inhaler/ MDPI) followed by cumulative doses (3 doses at 20 min intervals, administered via spacer) of placebo at 1h, 12h and 24h of dosing.
  Interventions: Drug: 400 microgrammes GSK961081

INTERVENTIONS:
Drug: 400 microgrammes GSK961081 — Inhaled GSK961081 administered via Dry Powder Inhaler.
  Arms: 1200 microgrammes GSK961081 and salbutamol; 1200 microgrammes of GSK961081 and ipratropium bromide; 1200 microgrammes of GSK961081 and placebo; 400 microgrammes GSK961081 and salbutamol
Drug: 1200 microgrammes GSK961081 — Inhaled GSK961081 adminisntered via dry powder inhaler.
  Arms: 1200 microgrammes GSK961081 and salbutamol; 1200 microgrammes of GSK961081 and ipratropium bromide; 400 microgrammes GSK961081 and ipratropium bromide; 400 microgrammes of GSK961081 and placebo

SUMMARY:
GSK961081 is a potent dual pharmacophore that demonstrates both antimuscarinic and beta-agonist pharmacology in preclinical studies, both pharmacologies being of long duration. If reproduced in man, GSK961081 has the potential to deliver a medicine that can be given once daily. The bronchodilatation after inhalation of single doses of GSK961081 alone and in the presence of the short acting beta agonist salbutamol and the short acting muscarinic antagonist, ipratropium bromide will be measured in this study. Any residual bronchodilatation post-inhalation of GSK961081 and demonstrated by addition of salbutamol or ipratropium bromide may provide an indirect assessment of the beta-agonist and antimuscarinic components of GSK961081

DETAILED DESCRIPTION:
GSK961081 is a potent dual pharmacophore that demonstrates both antimuscarinic and beta-agonist pharmacology in preclinical studies, both pharmacologies being of long duration. If reproduced in man, GSK961081 has the potential to deliver a medicine that can be given once daily. The bronchodilatation after inhalation of single doses of GSK961081 alone and in the presence of the short acting beta agonist salbutamol and the short acting muscarinic antagonist, ipratropium bromide will be measured in this study. Any residual bronchodilatation post-inhalation of GSK961081 and demonstrated by addition of salbutamol or ipratropium bromide may provide an indirect assessment of the beta-agonist and antimuscarinic components of GSK961081

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female (of non-child bearing potential) ≥ 40 years of age and ≤ 75 years of age.
* Non- child bearing potential is defined as physiologically incapable of becoming pregnant, including females who are post-menopausal (more than 2 years without menses with appropriate clinical history i.e. age, history of vasomotor symptoms-estradiol and FSH levels may be checked if indicated) and females who are surgically sterile (hysterectomy, tubal ligation or bilateral oophorectomy).
* Subject diagnosed with COPD in accordance with ATS/ERS guidelines (as per protocol).
* Subject is a smoker or an ex-smoker with a history of at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent)
* Subject has FEV1/FVC < 0.7 post-bronchodilator (salbutamol)
* Subject has FEV1 < 80 % of predicted normal for height, age, gender after inhalation of salbutamol
* Response to ipatropium bromide defined as:
* Either an increase in FEV1 of > 12 % and > 150 mL within 2 hours following inhalation of 80 µg ipratopium bromide (Atrovent MDI via spacer) at the screening visit
* Or: a documented increase in FEV1 of >12 % and > 150 mL within 2 hours following inhalation of 80 µg ipratopium bromide within 6 months of screening and an increase in FEV1 of > 6 % and > 100 mL within 2h following inhalation of 80 µg ipratopium bromide (Atrovent MDI via spacer) at the screening visit (in order to allow for potential fluctuations in the response to ipratropium bromide in patients known to be responders to ipratropium bromide)
* Response to salbutamol defined as:
* Either an increase in FEV1 of > 12 % and > 150 mL within 2 hours following inhalation of 400 µg salbutamol MDI (via spacer) at the screening visit
* Or: a documented increase in FEV1 of >12 % and > 150 mL within 2 hours following inhalation of 400 µg salbutamol MDI within 6 months of screening and an increase in FEV1 of > 6 % and >100 mL within 2h following inhalation of 400 µg salbutamol MDI (via spacer) at the screening visit (in order to allow for potential fluctuations in the response to salbutamol in patients known to be responders to salbutamol)
* Body mass index (BMI) within the range 18-35 kg/m2
* Subject is able and willing to give written informed consent to take part in the study.
* Subject is available to complete all study assessments

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the Investigator and medical monitor may affect the outcome of the study or the safety of the subject
* Subjects with clinically relevant findings on laboratory safety tests. Subjects with laboratory values outside the reference range may be include in the study if the Investigator and medical monitor agree that these findings would not put the subject at risk or interfere with the objectives of the study
* Women who are pregnant or lactating
* An unwillingness of subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or tubal ligation if the woman could become pregnant from the time of the first dose study medication until 90 days post-dose
* The subject has a positive urine drugs of abuse screen. A minimum list of drugs that will be screened for include amphetamines, barbituates, cocaine, opiates, cannabinoids and benzodiazepines.
* A history, or suspected history, of alcohol abuse within the 6 months before the screening visit.
* A positive test for hepatitis C antibody, hepatitis B surface antigen, or HIV.
* The subject has participated in a clinical study with another New Chemical Entity within the past 2 months or participated in a clinical study with any other drug during the previous month.
* The subject has donated a unit of blood within the 56 days of dosing or intends to donate within 56 days after completing the study.
* Subject has an FEV1 < 40 % of predicted for age, height and gender after inhalation of salbutamol.
* The subject has a diagnosis of active tuberculosis, lung cancer, sarcoidosis, bronchiectasis, lung fibrosis, pulmonary hypertension or with a primary diagnosis of asthma
* The subject has a known allergy or hypersensitivity to ipratropium bromide, salbutamol, or lactose
* A subject in whom ipratropium bromide or salbutamol is contraindicated
* Subjects with lung volume reduction surgery within 12 months of screening
* Poorly controlled COPD defined as:
* Either: acute worsening of COPD that is managed by the subject at home by treatment with increased corticosteroids or antibiotics in the 6 weeks before screening
* Or: more than 2 exacerbations in the previous 12 months before screening that required a course of oral steroids or antibiotics, and/or required hospitalisation
* Subject has had a respiratory tract infection in the 4 weeks before screening
* Subject requires treatment with inhaled cromolyn sodium, theophyline, oral ß2- agonists, nebulised anticholinergics or leukotriene antagonists
* Subject is unable to abstain from long acting ß2-agonist from 72 hours before screening and throughout the dosing period
* Subject is unable to abstain from tiotropium bromide from 28 days before screening and throughout the dosing period
* Subject is predicted to be unable to abstain from short acting inhaled ß2-agonists or short acting antimuscarinics for 6 hours before screening and for 6 hours before dosing with GSK961081 until all post-dose lung function tests have been completed for a given study day.
* Subject has received oral corticosteroids within the 6 weeks before screening
* Subject is receiving > 1000 µg FP (or equivalent) a day of inhaled corticosteroid or has changed dose within the 6 weeks before screening or is predicted not to be able to maintain a constant dose during the study
* Subject is receiving oxygen therapy or nocturnal positive pressure treatment
* Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the study investigator would prevent use of an inhaled anticholinergic
* The subject is unable to use the dosing devices (MDPI/ MDI/ spacer) correctly.
* Subject with carcinoma that has not been in complete remission for at least 5 years (with the exception of carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma if the subject is considered cured)
* A history of congestive heart failure, coronary insufficiency or cardiac arrhythmia or a finding on screening 24h Holter monitor that would contraindicate the subject's participation in the study
* 12- lead ECG abnormality which is either clinically significant or may interfere with QTc measurement or QTc > 450 msec or PR interval outside the range 120 to 220 msec.
* A supine mean heart rate outside the range 40-90 bpm at screening.
* Persistently elevated supine blood pressure higher than 160/95 at screening.
* Subject is receiving a high-dose diuretic and/ or ß2-adrenergic antagonist
* Subject has a serum potassium level below the reference range at screening.
* Inability to understand the protocol requirements, instructions and study-related restrictions; the nature, scope and possible consequences of the study.
* Unlikely to complete the study; e.g., uncooperative attitude, inability to return for follow-up visits.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-04-01; Primary Completion 2008-10-01 (Actual); Study Completion 2008-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Wellington, New Zealand
- Thailand (2):
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Norris V, Ambery C. Bronchodilation and safety of supratherapeutic doses of salbutamol or ipratropium bromide added to single dose GSK961081 in patients with moderate to severe COPD. Pulm Pharmacol Ther. 2013 Oct;26(5):574-80. doi: 10.1016/j.pupt.2013.03.009. Epub 2013 Mar 21. PMID 23524017
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAB110123 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 25Apr2008 to 19Oct2008 across two centers in Thailand and one center each in the United Kingdom and New Zealand. A total of 45 participants were planned to be enrolled.
Pre-assignment Details: A total of 44 participants were screened over period of 28 days and were enrolled in the study.
Groups:
- Total Population: Eligible participants received GSK961981 400 micrograms (mcg) and 1200 mcg metered Dry Powder Inhaler/ MDPI) followed by cumulative doses (3x 200 mcg at 0 min intervals, administered via spacer) of salbutamol at 1hour (h), 12h and 24h of dosing during first and second treatment periods, respectively. Eligible participants received GSK961981 400 mcg and 1200 mcg followed by cumulative doses (20 mcg , 20 mcg and 40 mcg at 20 minutes intervals, administered via spacer) of ipratropium bromide at 1h, 12h and 24h of dosing during third and forth treatment period, respectively. Eligible participants received GSK961981 400 mcg and 1200 mcg followed by cumulative doses (3 doses at 20 minutes intervals, administered via spacer) of Placebo at 1h, 12h and 24h of dosing during fifth and sixth treatment period, respectively.
Period: Period 1
Arm/Group | Total Population
Started | 44
Completed | 41
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Period: Period 2
Arm/Group | Total Population
Started | 41
Completed | 41
Not Completed | 0
Period: Period 3
Arm/Group | Total Population
Started | 41
Completed | 39
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Period: Period 4
Arm/Group | Total Population
Started | 39
Completed | 38
Not Completed | 1
Not completed — Adverse Event | 1
Period: Period 5
Arm/Group | Total Population
Started | 38
Completed | 38
Not Completed | 0
Period: Period 6
Arm/Group | Total Population
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects population included all participants who received at least one dose of the study drug.
Arm/Group | Total Population
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 63.1 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - South East Asian Heritage | 22
  Native Hawaiian or other Pacific Islander | 1
  White - White/Caucasian/European Heritage | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change in Forced Expiratory Volume in One Second (FEV1) From Baseline (Pre-dose on Day 1) in Combination With Short Acting Bronchodialator (Salbutamol or Ipratropium Bromide) at 1h,12h and 24h.
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second as measured by spirometry. Adjusted mean has been presented as least square (LS) mean.
Time Frame: Baseline (pre-dose on Day 1), 1h, 12h, and 24h on Day 1
Population: Modified per protocol population included the participants who received at least one dose of the study drug where major deviations from the protocol had not occurred. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- GSK961081 400 mg Plus SAL: Eligible participants received 400 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (3x 200 mcg at 20 min intervals, administered via spacer) of salbutamol at 1h, 12h and 24h of dosing.
- GSK961081 1200 mg Plus SAL: Eligible participants received 1200 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (3x 200 mcg at 20 min intervals, administered via spacer) of salbutamol at 1h, 12h and 24h of dosing.
- GSK961081 400 mg Plus IPR: Eligible participants received 400 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (20 mcg, 20 mcg and 40 microgrammes at 20 min intervals, administered via spacer) of ipratropium bromide at 1h, 12h and 24h of dosing.
- GSK961081 1200 mg Plus IPR: Eligible participants received 1200 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (20 mcg, 20 mcg, and 40 mcg at 20 min intervals, administered via spacer) of ipratropium bromide at 1h, 12h and 24h of dosing.
- GSK961081 400 mg Plus Placebo: Eligible participants received 400 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (3 doses at 20 min intervals, administered via spacer) of placebo at 1h, 12h and 24h of dosing.
- GSK961081 1200 mg Plus Placebo: Eligible participants received 1200 mcg of GSK961081 single-dose (via DISKUS MDPI) followed by cumulative doses (3 doses at 20 min intervals, administered via spacer) of placebo at 1h, 12h and 24h of dosing.
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Liters
  1 hour: number analyzed (Participants) | 39 | 41 | 40 | 40 | 37 | 37
  1 hour | 0.111 (0.0146) | 0.113 (0.0142) | 0.087 (0.0144) | 0.111 (0.0144) | 0.072 (0.0144) | 0.094 (0.0149)
  12 hour: number analyzed (Participants) | 39 | 40 | 40 | 40 | 40 | 38
  12 hour | 0.141 (0.0173) | 0.134 (0.0170) | 0.127 (0.0170) | 0.098 (0.0171) | 0.002 (0.0170) | 0.043 (0.0174)
  24 hour: number analyzed (Participants) | 39 | 40 | 41 | 39 | 40 | 37
  24 hour | 0.161 (0.0166) | 0.175 (0.0163) | 0.179 (0.0162) | 0.172 (0.0166) | 0.039 (0.0163) | 0.049 (0.0169)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo' at 1 hour; Test type: Superiority or Other; p = 0.020, Mix model; Mean Difference (Final Values) = 0.039, 90% CI 2-sided [0.008 to 0.069], Standard Error of Mean 0.0187
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p < 0.001, Mix model; Mean Difference (Final Values) = 0.139, 90% CI 2-sided [0.101 to 0.176], Standard Error of Mean 0.0227
Statistical Analysis 3: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p < 0.001, Mix model; Median Difference (Final Values) = 0.123, 90% CI 2-sided [0.087 to 0.158], Standard Error of Mean 0.0217
Statistical Analysis 4: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.220, Mix model; Mean Difference (Final Values) = 0.014, 90% CI 2-sided [-0.016 to 0.045], Standard Error of Mean 0.0185
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p < 0.001, Mix model; Mean Difference (Final Values) = 0.124, 90% CI 2-sided [0.087 to 0.161], Standard Error of Mean 0.0225
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p < 0.001, Mix model; Median Difference (Final Values) = 0.141, 90% CI 2-sided [0.105 to 0.176], Standard Error of Mean 0.0214
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.155, Mix model; Mean Difference (Final Values) = 0.019, 90% CI 2-sided [-0.012 to 0.050], Standard Error of Mean 0.0188
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p < 0.001, Mix model; Mean Difference (Final Values) = 0.091, 90% CI 2-sided [0.053 to 0.129], Standard Error of Mean 0.0229
Statistical Analysis 9: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p < 0.001, Mix model; Mean Difference (Final Values) = 0.126, 90% CI 2-sided [0.090 to 0.162], Standard Error of Mean 0.0220
Statistical Analysis 10: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.188, Mix model; Mean Difference (Final Values) = 0.017, 90% CI 2-sided [-0.015 to 0.048], Standard Error of Mean 0.0190
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p = 0.009, Mix model; Mean Difference (Final Values) = 0.055, 90% CI 2-sided [0.017 to 0.093], Standard Error of Mean 0.0230
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p < 0.001, Mix model; Mean Difference (Final Values) = 0.122, 90% CI 2-sided [0.086 to 0.159], Standard Error of Mean 0.0222

2. Secondary Outcome: Maximal Change in Forced Vital Capacity (FVC) in One Second From Pre-dose in Combination With Short Acting Bronchodialator (Salbutamol or Ipratropium Bromide) at 1h, 12h and 24h.
Description: FVC is defined as the amount of air that can be forcibly exhaled from the lungs after a maximum inspiration as measured by spirometry. Adjusted mean has been presented as least square (LS) mean.
Time Frame: Baseline (Pre-dose on Day 1), 1h, 12h, and 24h on Day 1
Population: Modified per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Liters
  1 hour: number analyzed (Participants) | 39 | 41 | 40 | 40 | 40 | 37
  1 hour | 0.169 (0.0460) | 0.281 (0.0449) | 0.167 (0.0454) | 0.207 (0.0454) | 0.234 (0.0454) | 0.229 (0.0472)
  12 hour: number analyzed (Participants) | 39 | 40 | 40 | 40 | 40 | 38
  12 hour | 0.160 (0.0380) | 0.182 (0.0375) | 0.188 (0.0375) | 0.223 (0.0375) | 0.068 (0.0375) | 0.088 (0.0385)
  24 hour: number analyzed (Participants) | 39 | 40 | 41 | 39 | 40 | 37
  24 hour | 0.247 (0.0398) | 0.205 (0.0392) | 0.279 (0.0388) | 0.214 (0.0397) | 0.179 (0.0393) | 0.113 (0.0407)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.856, Mix model; Mean Difference (Final Values) = -0.066, 90% CI 2-sided [-0.168 to 0.036], Standard Error of Mean 0.0616
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p = 0.033, Mix model; Mean Difference (Final Values) = 0.092, 90% CI 2-sided [0.010 to 0.174], Standard Error of Mean 0.0496
Statistical Analysis 3: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p = 0.099, Mix model; Mean Difference (Final Values) = 0.068, 90% CI 2-sided [-0.019 to 0.154], Standard Error of Mean 0.0523
Statistical Analysis 4: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.862, Mix model; Mean Difference (Final Values) = -0.067, 90% CI 2-sided [-0.168 to 0.034], Standard Error of Mean 0.0612
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p = 0.008, Mix model; Mean Difference (Final Values) = 0.120, 90% CI 2-sided [0.039 to 0.201], Standard Error of Mean 0.0493
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p = 0.027, Mix model; Mean Difference (Final Values) = 0.100, 90% CI 2-sided [0.015 to 0.185], Standard Error of Mean 0.0516
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.200, Mix model; Mean Difference (Final Values) = 0.052, 90% CI 2-sided [-0.050 to 0.155], Standard Error of Mean 0.0621
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus that due to GSK961081 1200 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p = 0.031, Mix model; Mean Difference (Final Values) = 0.094, 90% CI 2-sided [0.011 to 0.177], Standard Error of Mean 0.0500
Statistical Analysis 9: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p = 0.043, Mix model; Mean Difference (Final Values) = 0.092, 90% CI 2-sided [0.004 to 0.179], Standard Error of Mean 0.0530
Statistical Analysis 10: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 1 hour; Test type: Superiority or Other; p = 0.637, Mix model; Mean Difference (Final Values) = -0.022, 90% CI 2-sided [-0.125 to 0.081], Standard Error of Mean 0.0625
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 12 hour; Test type: Superiority or Other; p = 0.004, Mix model; Mean Difference (Final Values) = 0.136, 90% CI 2-sided [0.053 to 0.218], Standard Error of Mean 0.0500
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo at 24 hour; Test type: Superiority or Other; p = 0.031, Mix model; Mean Difference (Final Values) = 0.100, 90% CI 2-sided [0.012 to 0.189], Standard Error of Mean 0.0534

3. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious AE (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Upto 82 days
Population: All subjects population
Measure: Number; unit: Participants
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
Participants
  Participants with any AE | 13 | 13 | 15 | 9 | 6 | 11
  Participants with any SAE | 0 | 1 | 1 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities of Potential Clinical Concern (PCC)
Description: The normal ranges of laboratory parameters were hemoglobin: 130-167 grams per deciliter (g/dL), platelets: 173-383 Giga per liter (GI/L), lymphocytes: 20.1-44.5 %, glucose: 3.8857-6.106 millimoles per liter (mmol/L), creatinine: 44.2-132.6 micromoles per liter (uM/L) , aspartate transaminases (AST): 12-32 international units per liter (IU/L), total bilirubin (TB): 4.275-25.65 uM/L and potassium: 3.4-4.7 mmol/L, respectively. Laboratory values recorded outside the normal range were considered of potential clinical concern (PCC).
Time Frame: Up to 42 days
Population: All subjects population
Measure: Number; unit: Participants
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
Participants
  Hemoglobin high | 0 | 1 | 0 | 0 | 0 | 0
  Platelets high | 0 | 1 | 0 | 0 | 0 | 0
  Platelets low | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes low | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Change From Baseline (Pre-dose on Day 1) in Systolic and Diastolic Blood Pressure up to 27 Hours
Description: Change from Baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was analyzed. Change from baseline is the difference in the blood pressure at the indicated time point minus the Baseline value.
Time Frame: Up to 27 hours post Day 1 dosing
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm of Hg)
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
Millimeters of mercury (mm of Hg)
  SBP, 1 hour(h) | -1.33 (12.321) | 3.10 (11.115) | 0.61 (10.703) | -1.73 (10.301) | -0.13 (12.096) | -0.33 (11.235)
  SBP, 2h: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 39
  SBP, 2h | -3.41 (10.918) | 1.22 (10.741) | 3.49 (7.919) | 2.33 (11.450) | 1.03 (8.195) | 1.31 (12.131)
  SBP, 4h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  SBP, 4h | -2.36 (8.963) | 4.20 (12.107) | 3.27 (9.680) | 2.68 (9.689) | 0.63 (10.947) | 2.38 (10.101)
  SBP, 9h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  SBP, 9h | -0.87 (12.064) | 3.08 (10.598) | 1.07 (10.900) | 2.71 (12.125) | 0.00 (9.748) | 2.95 (12.237)
  SBP, 12h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  SBP, 12h | -3.49 (11.850) | 2.08 (15.895) | -0.46 (11.145) | 0.32 (12.445) | -1.95 (11.618) | -0.51 (10.450)
  SBP, 13h: number analyzed (Participants) | 37 | 39 | 41 | 41 | 40 | 38
  SBP, 13h | -5.62 (11.947) | 3.46 (13.742) | 1.05 (11.866) | 2.27 (13.808) | 3.45 (15.591) | 2.21 (9.935)
  SBP, 24h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  SBP, 24h | -3.31 (12.092) | 4.65 (10.843) | 1.41 (11.469) | 2.56 (12.616) | -1.50 (10.627) | 1.68 (10.547)
  SBP, 25h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 37
  SBP, 25h | -3.38 (11.679) | 4.05 (14.022) | 2.32 (13.083) | 2.44 (9.453) | -0.10 (12.349) | 1.49 (11.428)
  SBP, 27h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  SBP, 27h | -5.59 (9.999) | 2.43 (11.670) | -3.24 (11.432) | -0.32 (12.875) | -3.25 (10.463) | -1.24 (10.899)
  DBP, 1h: number analyzed (Participants) | 39 | 41 | 40 | 41 | 40 | 39
  DBP, 1h | -1.59 (6.754) | -1.41 (6.340) | 1.25 (8.002) | -2.66 (6.814) | 0.55 (6.737) | -2.21 (8.594)
  DBP, 2h: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 39
  DBP, 2h | -4.15 (7.744) | -2.27 (7.871) | 0.07 (7.438) | 0.48 (6.939) | -1.48 (6.473) | -1.05 (7.189)
  DBP, 4h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  DBP, 4h | -0.26 (6.332) | 1.23 (6.078) | 1.24 (6.689) | 0.12 (8.134) | 1.38 (8.350) | 1.54 (6.353)
  DBP, 9h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  DBP, 9h | -1.59 (7.923) | 0.03 (7.882) | -1.73 (7.820) | -0.34 (9.175) | 0.28 (6.373) | -0.79 (8.581)
  DBP, 12h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  DBP, 12h | -3.18 (8.742) | -1.25 (7.655) | -2.68 (8.329) | -0.90 (7.605) | -3.05 (7.414) | -0.51 (7.026)
  DBP, 13h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  DBP, 13h | -4.19 (11.638) | -1.97 (7.856) | -0.56 (8.152) | -0.39 (7.602) | 0.85 (9.670) | -0.34 (8.380)
  DBP, 24h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  DBP, 24h | -0.95 (6.411) | 3.13 (8.624) | 0.37 (5.634) | 2.32 (7.932) | -0.23 (6.799) | -0.58 (7.310)
  DBP, 25h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 37
  DBP, 25h | -2.26 (6.976) | 0.75 (7.171) | 1.24 (8.166) | 1.49 (8.474) | 0.78 (5.753) | 2.22 (7.536)
  DBP, 27h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  DBP, 27h | -3.28 (7.229) | -0.03 (8.192) | -2.51 (7.871) | -1.12 (7.541) | -3.35 (9.270) | -1.55 (7.202)

6. Secondary Outcome: Mean Change From Baseline (Pre-dose on Day 1) in Heart Rate Over 27 Hours
Description: Heart rate was considered as a measure of vital sign. Change from baseline is the difference in the blood pressure at the indicated time point minus the Baseline value.
Time Frame: Up to 27 hours post Day 1 dosing
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
Beats per minute
  1h | -2.56 (10.246) | -1.37 (8.546) | -3.90 (7.761) | -2.27 (7.099) | -3.55 (9.047) | -3.10 (6.585)
  1h 15 minutes: number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 38
  1h 15 minutes | -0.95 (8.712) | -0.46 (7.328) | -2.80 (7.118) | -0.15 (6.624) | -4.03 (7.540) | -1.74 (5.915)
  1h 35 minutes: number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 38
  1h 35 minutes | -0.03 (8.481) | 1.51 (7.166) | -2.34 (7.275) | -0.98 (5.943) | -3.63 (6.717) | -2.36 (6.098)
  1h 55 minutes: number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 38
  1h 55 minutes | 3.21 (9.359) | 4.54 (7.246) | -3.46 (7.232) | -0.39 (6.629) | -3.63 (6.636) | -2.21 (6.420)
  4h: number analyzed (Participants) | 38 | 40 | 41 | 41 | 40 | 39
  4h | -0.71 (11.094) | 1.13 (6.501) | -3.59 (9.389) | -1.78 (6.031) | -4.75 (6.636) | -3.97 (7.069)
  9h: number analyzed (Participants) | 39 | 39 | 41 | 41 | 40 | 39
  9h | 1.92 (6.247) | 2.97 (6.815) | -1.66 (7.529) | 1.37 (7.569) | -0.70 (8.879) | 0.28 (7.215)
  12h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 39
  12h | 1.95 (7.567) | 3.65 (8.469) | 1.46 (8.521) | 2.83 (7.752) | 2.68 (8.689) | 1.87 (6.993)
  12h 15 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  12h 15 minutes | 3.95 (7.729) | 5.35 (7.608) | 1.83 (6.364) | 4.10 (7.612) | 1.80 (6.992) | 2.05 (8.220)
  12h 35 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  12h 35 minutes | 4.97 (7.741) | 6.90 (7.558) | 1.51 (6.856) | 3.41 (8.465) | 2.28 (6.520) | 1.29 (6.534)
  12h 55 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  12h 55 minutes | 5.79 (8.694) | 6.50 (8.124) | 1.07 (7.424) | 1.90 (7.671) | 0.98 (7.416) | 1.37 (8.065)
  24h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  24h | -2.36 (8.142) | -1.08 (7.145) | -3.24 (5.267) | -1.85 (7.189) | -3.63 (8.079) | -4.55 (7.576)
  24h 15 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  24h 15 minutes | -1.49 (8.705) | -1.60 (7.938) | -0.83 (7.297) | -0.98 (7.666) | -2.95 (6.972) | -4.03 (8.284)
  24h 35 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  24h 35 minutes | 0.23 (8.806) | 0.53 (7.990) | -2.93 (6.218) | -1.02 (6.901) | -4.48 (6.361) | -4.63 (6.724)
  24h 55 minutes: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  24h 55 minutes | 1.05 (8.617) | 0.83 (8.650) | -2.46 (9.223) | -2.05 (6.488) | -4.13 (7.198) | -4.21 (7.037)
  27h: number analyzed (Participants) | 39 | 40 | 41 | 41 | 40 | 38
  27h | 6.74 (9.402) | 6.38 (9.440) | 1.17 (9.132) | 4.44 (9.394) | 2.05 (7.968) | 2.68 (8.817)

7. Secondary Outcome: Number of Participants With Maximum Change From Baseline 12-LED Electrocardiogram (ECG) Findings
Description: Analysis QTc interval of ECG was performed by Bazett's formula (QTc B) and Fridericia's correction (QTc F). Number of participants with abnormal ECG findings were recorded. Any participant with QTc(B) or QTc(F) >500 milliseconds (msec) or uncorrected QT >600 msec (machine or manual over read) was withdrawn from the study. Participants that had right bundle branch block with QTc(B) or QTc(F) >530 msec were also withdrawn from the study.
Time Frame: From dosing until 24h post-dose.
Population: All subjects population
Measure: Number; unit: Participants
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
Participants
  QTcB, <=30 msec | 26 | 31 | 35 | 33 | 36 | 31
  QTcB, >30 to <= 59 msec | 12 | 9 | 6 | 7 | 3 | 6
  QTcB, >=60 msec | 1 | 1 | 0 | 1 | 1 | 2
  QTcF, <=30 msec | 34 | 31 | 37 | 36 | 36 | 35
  QTcF, >30 to <= 59 msec | 5 | 9 | 2 | 4 | 4 | 2
  QTcF, >=60 msec | 0 | 1 | 2 | 1 | 0 | 2

8. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in QTc (F) in Supine Position From 0 to 4 Hours After Dosing
Description: Analysis of QT (F) interval during ECG (taken in supine position) was performed using Fridericia's method. Change from baseline is the value at indicated time point minus the value at Baseline. Adjusted means are considered as least square (LS) mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h)
Population: Modified per protocol population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
msec | 14.34 (1.865) | 14.98 (1.827) | 12.31 (1.824) | 11.99 (1.839) | 10.60 (1.844) | 13.22 (1.890)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 3.747, 95% CI 2-sided [-0.547 to 8.041], Standard Error of Mean 2.1768
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.712, 95% CI 2-sided [-2.521 to 5.944], Standard Error of Mean 2.1453
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.755, 95% CI 2-sided [-2.559 to 6.069], Standard Error of Mean 2.1869
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.231, 95% CI 2-sided [-5.565 to 3.103], Standard Error of Mean 2.1970

9. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in QTc (F) in Supine Position From 0 to 27 Hours After Dosing
Description: Analysis of Q T (F) interval during ECG (taken in supine position) was performed using Fridericia's method. Change from baseline is the value at indicated time point minus the value at Baseline. Adjusted means are considered as LS mean values while presenting the data .
Time Frame: From dosing until 27 hours (0-27h)
Population: Modified per protocol population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
msec | 19.70 (2.152) | 19.53 (2.104) | 17.41 (2.100) | 17.45 (2.119) | 15.14 (2.125) | 18.60 (2.184)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo over 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 4.558, 95% CI 2-sided [-0.781 to 9.897], Standard Error of Mean 2.7064
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo over 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 2.266, 95% CI 2-sided [-2.999 to 7.532], Standard Error of Mean 2.6691
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo over 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.930, 95% CI 2-sided [-4.429 to 6.290], Standard Error of Mean 2.7170
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo over 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.152, 95% CI 2-sided [-6.539 to 4.236], Standard Error of Mean 2.7310

10. Secondary Outcome: Weighted Mean Change From Baseline (Pre-dose on Day 1) in QTc(F) in Supine Position From 0 to 4 Hours
Description: Analysis of QT(F) interval during ECG (taken in supine position) was performed using Fridericia's method. Change from baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h)
Population: Modified per protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: msec
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 37
msec | 5.42 (1.565) | 7.53 (1.536) | 4.59 (1.535) | 6.23 (1.546) | 4.17 (1.549) | 8.18 (1.597)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.249, 95% CI 2-sided [-2.069 to 4.566], Standard Error of Mean 1.6816
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.418, 95% CI 2-sided [-2.850 to 3.687], Standard Error of Mean 1.6565
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.650, 95% CI 2-sided [-4.013 to 2.714], Standard Error of Mean 1.7050
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo over 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.949, 95% CI 2-sided [-5.325 to 1.427], Standard Error of Mean 1.7112

11. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in QTc(B) in Supine Position From 0 to 4 Hours and 0 to 27 Hours
Description: Analysis of QT (B) interval during ECG (taken in supine position) was performed using Bazett's method. Change from baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data .
Time Frame: From dosing until 4 hours (0-4h) and 27 hours (0-27h)
Population: Modified Per Protocol population.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
msec
  0-4 hours | 16.70 (2.078) | 19.51 (2.035) | 9.19 (2.033) | 10.77 (2.047) | 6.50 (2.054) | 11.65 (2.109)
  0-27 hours | 24.17 (2.390) | 25.88 (2.339) | 17.33 (2.337) | 17.83 (2.353) | 12.94 (2.362) | 19.91 (2.429)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 10.198, 95% CI 2-sided [5.258 to 15.139], Standard Error of Mean 2.5039
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 2.686, 95% CI 2-sided [-2.195 to 7.567], Standard Error of Mean 2.4738
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 7.854, 95% CI 2-sided [2.883 to 12.825], Standard Error of Mean 2.5196
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.884, 95% CI 2-sided [-5.864 to 4.097], Standard Error of Mean 2.5244
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 11.227, 95% CI 2-sided [5.352 to 17.103], Standard Error of Mean 2.9782
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 4.390, 95% CI 2-sided [-1.418 to 10.197], Standard Error of Mean 2.9434
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 5.975, 95% CI 2-sided [0.065 to 11.886], Standard Error of Mean 2.9958
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -2.083, 95% CI 2-sided [-8.006 to 3.840], Standard Error of Mean 3.0023

12. Secondary Outcome: Weighted Mean Change From Baseline (Pre-dose on Day 1) in QTc(B) in Supine Position From 0 to 4 Hours
Description: Analysis of QT (B) interval during ECG (taken in supine position) was performed using Bazett's method. Change from baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h)
Population: Modified Per Protocol population.
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 37
msec | 5.27 (1.569) | 9.08 (1.542) | 0.08 (1.542) | 4.44 (1.550) | 0.07 (1.555) | 6.12 (1.602)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 5.200, 95% CI 2-sided [1.857 to 8.542], Standard Error of Mean 1.6941
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-3.294 to 3.307], Standard Error of Mean 1.6727
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 2.956, 95% CI 2-sided [-0.433 to 6.345], Standard Error of Mean 1.7178
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.683, 95% CI 2-sided [-5.076 to 1.711], Standard Error of Mean 1.7199

13. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in Supine Heart Rate From 0 to 4 Hours and From 0 to 27 Hours.
Description: Heart rate was measured in supine position. Change from baseline is the value at indicated time point minus the value at Baseline. Adjusted means are considered as LS mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h) and until 27 hours (0-27 h)
Population: Modified Per Protocol population.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Beats per minute
  0-4 h | 7.51 (1.125) | 7.90 (1.099) | 2.18 (1.097) | 3.17 (1.109) | 0.92 (1.110) | 0.92 (1.139)
  0-27 h | 13.33 (1.011) | 12.92 (0.988) | 9.49 (0.987) | 10.28 (0.998) | 9.21 (0.998) | 8.66 (1.024)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 6.588, 95% CI 2-sided [3.839 to 9.336], Standard Error of Mean 1.3932
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.255, 95% CI 2-sided [-1.453 to 3.962], Standard Error of Mean 1.3725
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 6.985, 95% CI 2-sided [4.231 to 9.738], Standard Error of Mean 1.3960
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 2.255, 95% CI 2-sided [-0.522 to 5.031], Standard Error of Mean 1.4077
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus maximal GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 4.121, 95% CI 2-sided [1.662 to 6.580], Standard Error of Mean 1.2464
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.280, 95% CI 2-sided [-2.142 to 2.703], Standard Error of Mean 1.2278
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 4.266, 95% CI 2-sided [1.802 to 6.729], Standard Error of Mean 1.2490
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.621, 95% CI 2-sided [-0.863 to 4.106], Standard Error of Mean 1.2593

14. Secondary Outcome: Weighted Mean Change From Baseline (Pre-dose on Day 1) in Heart Rate in Supine Position From 0 to 4 Hours
Description: Heart rate was recorded in supine position. Change from baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h)
Population: Modified Per Protocol population. Data is presented for the participants available at the time of assessment.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 37
Beats per minute | 0.52 (0.729) | 1.77 (0.713) | -2.93 (0.714) | -1.27 (0.720) | -3.57 (0.721) | -2.21 (0.745)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 4.094, 95% CI 2-sided [2.456 to 5.732], Standard Error of Mean 0.8300
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.646, 95% CI 2-sided [-0.967 to 2.258], Standard Error of Mean 0.8172
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 3.980, 95% CI 2-sided [2.324 to 5.636], Standard Error of Mean 0.8395
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.934, 95% CI 2-sided [-0.735 to 2.603], Standard Error of Mean 0.8460

15. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in Supine Systolic Blood Pressure (SBP) Over 4 and 27 Hours and Weighted Mean Change From Baseline in Supine SBP Over 4 Hours
Description: Systolic blood pressure (SBP) values were recorded in supine position. Change from baseline is the value at indicated time point minus the value at Baseline. Adjusted or maximum change/ (MC) and weighted mean change (WMC) are considered as LS mean change values while presenting the data.
Time Frame: 0-4h and 0-27h for maximum change and 0-4 h for weighted mean change
Population: Modified Per Protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Millimeters of mercury
  MC from BL,SBP,0-4h | 5.61 (1.452) | 8.06 (1.409) | 8.05 (1.394) | 5.55 (1.414) | 7.45 (1.412) | 7.74 (1.448)
  MC from BL,SBP,0-27h | 10.89 (1.530) | 15.93 (1.488) | 14.08 (1.477) | 12.87 (1.495) | 14.16 (1.493) | 14.10 (1.527)
  WMC from BL SBP,0-4h: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 37
  WMC from BL SBP,0-4h | -0.34 (1.103) | 0.92 (1.071) | 2.24 (1.063) | 0.10 (1.076) | 1.06 (1.075) | 0.82 (1.113)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.836, 95% CI 2-sided [-5.420 to 1.748], Standard Error of Mean 1.8168
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.599, 95% CI 2-sided [-2.914 to 4.113], Standard Error of Mean 1.7809
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.324, 95% CI 2-sided [-3.261 to 3.909], Standard Error of Mean 1.8174
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -2.182, 95% CI 2-sided [-5.781 to 1.416], Standard Error of Mean 1.8242
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -3.266, 95% CI 2-sided [-6.762 to 0.230], Standard Error of Mean 1.7723
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.077, 95% CI 2-sided [-3.502 to 3.348], Standard Error of Mean 1.7361
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.827, 95% CI 2-sided [-1.673 to 5.327], Standard Error of Mean 1.7743
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.232, 95% CI 2-sided [-4.743 to 2.279], Standard Error of Mean 1.7800
Statistical Analysis 9: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -1.394, 95% CI 2-sided [-3.976 to 1.187], Standard Error of Mean 1.3084
Statistical Analysis 10: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 1.181, 95% CI 2-sided [-1.348 to 3.710], Standard Error of Mean 1.2819
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [-2.498 to 2.710], Standard Error of Mean 1.3201
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.713, 95% CI 2-sided [-3.325 to 1.899], Standard Error of Mean 1.3241

16. Secondary Outcome: Minimum Change From Baseline (Pre-dose on Day 1) in Supine Diastolic Blood Pressure (DBP) Over 4 and 27 Hours and Weighted Mean Change From Baseline in Supine DBP Over 4 Hours
Description: Diastolic blood pressure (DBP) values were recorded in supine position. Change from baseline is the value at indicated time point minus the value at Baseline. Adjusted or maximum change/(MC) and weighted mean change (WMC) are considered as LS mean change values while presenting the data .
Time Frame: 0-4h and 0-27h for maximum change and 0-4 h for weighted mean change
Population: Modified Per Protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Millimeters of mercury
  MC from BL, DBP, 0-4h | -5.53 (0.971) | -5.76 (0.946) | -3.26 (0.942) | -5.49 (0.954) | -4.96 (0.954) | -4.42 (0.979)
  MC from BL, DBP, 0-27h | -10.04 (0.953) | -9.20 (0.930) | -9.12 (0.928) | -8.72 (0.938) | -9.66 (0.938) | -9.18 (0.959)
  WMC from BL, DBP, 0-4h: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 37
  WMC from BL, DBP, 0-4h | -1.30 (0.733) | -1.25 (0.715) | 0.75 (0.713) | -0.80 (0.721) | -0.12 (0.721) | -0.44 (0.747)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.561, 95% CI 2-sided [-2.997 to 1.876], Standard Error of Mean 1.2351
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 1.705, 95% CI 2-sided [-0.687 to 4.097], Standard Error of Mean 1.2125
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.337, 95% CI 2-sided [-3.771 to 1.098], Standard Error of Mean 1.2341
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -1.067, 95% CI 2-sided [-3.516 to 1.382], Standard Error of Mean 1.2416
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.376, 95% CI 2-sided [-2.545 to 1.794], Standard Error of Mean 1.0997
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.540, 95% CI 2-sided [-1.588 to 2.668], Standard Error of Mean 1.0786
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.016, 95% CI 2-sided [-2.185 to 2.154], Standard Error of Mean 1.0999
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.466, 95% CI 2-sided [-1.715 to 2.648], Standard Error of Mean 1.1058
Statistical Analysis 9: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -1.180, 95% CI 2-sided [-2.918 to 0.559], Standard Error of Mean 0.8810
Statistical Analysis 10: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.876, 95% CI 2-sided [-0.829 to 2.582], Standard Error of Mean 0.8644
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.809, 95% CI 2-sided [-2.561 to 0.944], Standard Error of Mean 0.8882
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.360, 95% CI 2-sided [-2.122 to 1.401], Standard Error of Mean 0.8929

17. Secondary Outcome: Maximum Change From Baseline (Pre-dose on Day 1) in Glucose Over 4 and 27 Hours and Weighted Mean Change From Baseline in Glucose Over 4 Hours
Description: Maximum change (MC) from Baseline (BL) and weighted mean change (WMC) from baseline in glucose (GLU) were analyzed. Change from Baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: 0-4h and 0-27h for maximum change and 0-4 h for weighted mean change
Population: Modified Per Protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per Liter
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Millimoles per Liter
  MC from BL, Glu, 0-4h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  MC from BL, Glu, 0-4h | 0.66 (0.186) | 0.53 (0.182) | 0.52 (0.182) | 0.53 (0.186) | 0.13 (0.184) | 0.22 (0.189)
  MC from BL, Glu, 0-27h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  MC from BL, Glu, 0-27h | 2.71 (0.236) | 2.13 (0.230) | 1.78 (0.230) | 1.87 (0.235) | 1.83 (0.232) | 1.30 (0.239)
  WMC from BL, Glu, 0-4h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 37
  WMC from BL, Glu, 0-4h | 0.02 (0.083) | 0.02 (0.081) | -0.12 (0.081) | -0.08 (0.082) | -0.29 (0.082) | 0.19 (0.085)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.530, 95% CI 2-sided [0.066 to 0.994], Standard Error of Mean 0.2352
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.388, 95% CI 2-sided [-0.069 to 0.846], Standard Error of Mean 0.2318
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.309, 95% CI 2-sided [-0.157 to 0.775], Standard Error of Mean 0.2363
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.309, 95% CI 2-sided [-0.163 to 0.780], Standard Error of Mean 0.2392
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.874, 95% CI 2-sided [0.262 to 1.485], Standard Error of Mean 0.3099
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-0.656 to 0.550], Standard Error of Mean 0.3056
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.829, 95% CI 2-sided [0.215 to 1.443], Standard Error of Mean 0.3112
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.567, 95% CI 2-sided [-0.054 to 1.189], Standard Error of Mean 0.3151
Statistical Analysis 9: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.312, 95% CI 2-sided [0.110 to 0.513], Standard Error of Mean 0.1021
Statistical Analysis 10: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus maximum GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [-0.025 to 0.372], Standard Error of Mean 0.1006
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.210, 95% CI 2-sided [0.006 to 0.414], Standard Error of Mean 0.1035
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [-0.103 to 0.311], Standard Error of Mean 0.1047

18. Secondary Outcome: Minimum Change From Baseline (Pre-dose on Day 1) in Potassium Over 4 and 27 Hours and Weighted Mean Change From Baseline in Potassium Over 4 Hours
Description: Maximum change (MC) from Baseline (BL) and weighted mean change (WMC) from baseline in potassium (K) were analyzed. Change from Baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: 0-4h and 0-27h for maximum change and 0-4 h for weighted mean change
Population: Modified Per Protocol population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per Liter
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
Millimoles per Liter
  MC from BL, K, 0-4h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  MC from BL, K, 0-4h | -0.42 (0.042) | -0.44 (0.041) | -0.25 (0.041) | -0.39 (0.042) | -0.25 (0.041) | -0.36 (0.042)
  MC from BL, K, 0-27h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  MC from BL, K, 0-27h | -0.53 (0.042) | -0.62 (0.040) | -0.42 (0.041) | -0.46 (0.041) | -0.37 (0.041) | -0.45 (0.042)
  WMC from BL, K, 0-4h: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 37
  WMC from BL, K, 0-4h | -0.18 (0.042) | -0.22 (0.040) | -0.06 (0.040) | -0.17 (0.041) | -0.07 (0.041) | -0.14 (0.042)
Statistical Analysis 1: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-0.276 to -0.078], Standard Error of Mean 0.0503
Statistical Analysis 2: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.096 to 0.097], Standard Error of Mean 0.0490
Statistical Analysis 3: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; SK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.076, 95% CI 2-sided [-0.174 to 0.022], Standard Error of Mean 0.0498
Statistical Analysis 4: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.128 to 0.072], Standard Error of Mean 0.0507
Statistical Analysis 5: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.166, 95% CI 2-sided [-0.263 to -0.069], Standard Error of Mean 0.0493
Statistical Analysis 6: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.057, 95% CI 2-sided [-0.152 to 0.038], Standard Error of Mean 0.0481
Statistical Analysis 7: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.171, 95% CI 2-sided [-0.267 to -0.075], Standard Error of Mean 0.0489
Statistical Analysis 8: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-27 hours; Test type: Superiority or Other; Mean Difference (Final Values) = -0.009, 95% CI 2-sided [-0.108 to 0.089], Standard Error of Mean 0.0498
Statistical Analysis 9: Comparison: GSK961081 400 mg Plus SAL vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus SAL versus GSK961081 400 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.108, 95% CI 2-sided [-0.211 to -0.005], Standard Error of Mean 0.0522
Statistical Analysis 10: Comparison: GSK961081 400 mg Plus IPR vs GSK961081 400 mg Plus Placebo; GSK961081 400 mcg Plus IPR versus GSK961081 400 mcg plus Placebo during 0-4 hours; Test type: Superiority or Other; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.087 to 0.114], Standard Error of Mean 0.0509
Statistical Analysis 11: Comparison: GSK961081 1200 mg Plus SAL vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus SAL GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.077, 95% CI 2-sided [-0.180 to 0.026], Standard Error of Mean 0.0520
Statistical Analysis 12: Comparison: GSK961081 1200 mg Plus IPR vs GSK961081 1200 mg Plus Placebo; GSK961081 1200 mcg Plus IPR versus GSK961081 1200 mcg plus Placebo during 0-4 hours (WMC); Test type: Superiority or Other; Mean Difference (Final Values) = -0.024, 95% CI 2-sided [-0.129 to 0.080], Standard Error of Mean 0.0529

19. Secondary Outcome: Time to Maximum Change From Baseline (Pre-dose on Day 1) for QTc(B), QTc(F), Heart Rate, Systolic BP, Glucose in Supine Position and Time to Minimum Change From Baseline for Potassium and Diastolic BP in Supine Position
Description: Analysis of QT (B) or QTc (F) interval during ECG (taken in supine position) was performed using Bazett's method and Fridericia's method, respectively. Heart rate, BP, potassium, and glucose were measured in supine body position. Change from baseline is the value at indicated time point minus the value at Baseline. Weighted means are considered as LS mean values while presenting the data.
Time Frame: From dosing until 4 hours (0-4h)
Population: Modified Per Protocol population. n=data is presented for the participants available at the time of assessment.
Measure: Median (Full Range); unit: hours
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 38
hours
  Heart rate: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
  Heart rate | 1.850 [0.88 to 4.0] | 1.850 [0.88 to 4.0] | 1.517 [0.87 to 3.98] | 1.517 [0.88 to 4.00] | 1.567 [0.88 to 3.98] | 1.567 [0.87 to 4.17]
  Systlic BP: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
  Systlic BP | 0.917 [0.87 to 3.98] | 2.100 [0.87 to 3.98] | 2.100 [0.90 to 3.98] | 2.100 [0.88 to 3.98] | 2.008 [0.87 to 3.98] | 3.008 [0.88 to 4.17]
  Diastolic BP: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
  Diastolic BP | 2.100 [0.87 to 3.97] | 1.967 [0.87 to 3.98] | 2.100 [0.87 to 4.02] | 0.933 [0.83 to 3.98] | 1.983 [0.88 to 3.97] | 0.925 [0.88 to 3.98]
  QTcF: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
  QTcF | 2.183 [0.83 to 3.98] | 2.100 [0.87 to 3.95] | 2.167 [0.83 to 4.03] | 2.100 [0.83 to 3.98] | 2.133 [0.63 to 4.00] | 2.117 [0.83 to 4.10]
  QTcB: number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 38
  QTcB | 2.100 [0.83 to 3.98] | 2.100 [0.87 to 3.95] | 2.100 [0.83 to 4.03] | 2.100 [0.83 to 3.98] | 2.100 [0.63 to 4.00] | 2.100 [0.83 to 4.10]
  Glucose: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  Glucose | 1.933 [0.92 to 4.00] | 1.950 [0.92 to 4.03] | 0.967 [0.90 to 4.00] | 0.967 [0.90 to 4.08] | 1.150 [0.92 to 4.03] | 0.967 [0.92 to 4.02]
  Potassium: number analyzed (Participants) | 39 | 41 | 41 | 39 | 40 | 38
  Potassium | 1.967 [0.92 to 4.43] | 1.933 [0.92 to 4.03] | 1.933 [0.92 to 4.00] | 1.950 [0.90 to 4.02] | 1.942 [0.88 to 4.05] | 1.933 [0.88 to 4.02]

20. Secondary Outcome: Area Under Plasma Concentration Time Curve (AUC) of GSK961081 to the Last Quantifiable Concentration
Description: AUC(0-t) is the area under plasma concentration time curve of GSK961081 to the last quantifiable concentration. This parameter was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. A large proportion of AUC(0-t) and Cmax values were reported as not countable (NC) at the GSK961081 400 micrograms (ug) dose level, therefore only limited summaries were calculated. Logarithmic transformed values are presented. AUC(0-t) imputed with 1/2 lowest observed AUC(0-t), where lowest AUC(0-t) was 56.46 hour picograms per milliliter (h*pg/mL).
Time Frame: Up to 82 days
Population: Pharmacokinetic (PK) population included participants in the 'All Subjects' population for whom a PK sample was obtained and analyzed following GSK961081 dosing. All participants were available at the time of analysis; however, for few participants, parameter cannot be derived because of non-quantifiable concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
h*pg/mL | NA (NA) — Not applicable due to insufficient data to derive summary measure | 233.93 (139.0) | NA (NA) — Not applicable due to insufficient data to derive summary measure | 216.22 (131.3) | NA (NA) — Not applicable due to insufficient data to derive summary measure | 229.51 (128.6)

21. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GSK961081 Over Period Determined Directly From the Concentration-time Data
Description: Cmax is the Maximum observed concentration of GSK961081 determined directly from the concentration-time data. A large proportion of Cmax values were reported as not countable (NC ) at the GSK961081 400 micrograms (ug) dose level, therefore only limited summaries were calculated. Logarithmic transformed values are presented. Cmax was imputed with 1/2 lowest limit of quantification (LLQ), where LLQ was 25 picograms per milliliter (pg/mL).
Time Frame: Up to 82 days
Population: PK population. All participants were present for analysis, however, there were few participants for whom parameter could not be derived because of non-quantifiable concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 39 | 41 | 41 | 41 | 40 | 39
pg/mL | 66.93 (55.0) | 169.05 (66.2) | 70.77 (54.8) | 153.59 (50.5) | 70.52 (60.9) | 176.92 (47.9)

22. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of GSK961081 Over Period Determined Directly From the Concentration-time Data
Description: Tmax is the time to maximum plasma concentration of GSK961081 over period determined directly from the concentration-time data
Time Frame: Up to 82 days
Population: PK population. All participants were present for the analysis; however, there were few participants for whom parameter could not be derived because of non-quantifiable concentrations. Data is presented for the participants available at the time of assessment.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 38 | 41 | 40 | 41 | 39 | 39
Hours | 0.920 [0.90 to 1.97] | 0.930 [0.90 to 2.08] | 0.925 [0.90 to 1.97] | 0.920 [0.90 to 1.97] | 0.920 [0.83 to 2.02] | 0.920 [0.83 to 1.93]

23. Secondary Outcome: Time to Last Quantifiable Plasma Concentration (Tlast) of GSK961081 Over Period Determined Directly From the Concentration-time Data
Description: Tlast is the time to last quantifiable plasma concentration of GSK961081 over period determined directly from the concentration-time data
Time Frame: Up to 82 days
Population: PK population. All participants were present for the analysis; however, there were few participants for whom parameter could not be derived because of non-quantifiable concentration. Data is presented for the participants available at the time of assessment.
Measure: Median (Full Range); unit: hours
Arm/Group | GSK961081 400 mg Plus SAL | GSK961081 1200 mg Plus SAL | GSK961081 400 mg Plus IPR | GSK961081 1200 mg Plus IPR | GSK961081 400 mg Plus Placebo | GSK961081 1200 mg Plus Placebo
Number analyzed (Participants) | 38 | 41 | 40 | 41 | 39 | 39
hours | 0.960 [0.90 to 4.02] | 2.000 [0.92 to 23.95] | 1.930 [0.92 to 11.95] | 3.920 [0.92 to 23.97] | 1.920 [0.83 to 4.00] | 2.050 [0.92 to 11.98]

ADVERSE EVENTS:
Time Frame: Up to 82 days
Description: All Subjects population included all participants who received at least one dose of the study drug.
Arm/Group | 400 Microgrammes GSK961081 and Salbutamol | 1200 Microgrammes GSK961081 and Salbutamol | 400 Microgrammes GSK961081 and Ipratropium Bromide | 1200 Microgrammes of GSK961081 and Ipratropium Bromide | 400 Microgrammes of GSK961081 and Placebo | 1200 Microgrammes of GSK961081 and Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/41 | 1/41 | 0/41 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 13/39 | 13/41 | 14/41 | 9/41 | 6/40 | 11/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 Microgrammes GSK961081 and Salbutamol (N=39) | 1200 Microgrammes GSK961081 and Salbutamol (N=41) | 400 Microgrammes GSK961081 and Ipratropium Bromide (N=41) | 1200 Microgrammes of GSK961081 and Ipratropium Bromide (N=41) | 400 Microgrammes of GSK961081 and Placebo (N=40) | 1200 Microgrammes of GSK961081 and Placebo (N=39)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 Microgrammes GSK961081 and Salbutamol (N=39) | 1200 Microgrammes GSK961081 and Salbutamol (N=41) | 400 Microgrammes GSK961081 and Ipratropium Bromide (N=41) | 1200 Microgrammes of GSK961081 and Ipratropium Bromide (N=41) | 400 Microgrammes of GSK961081 and Placebo (N=40) | 1200 Microgrammes of GSK961081 and Placebo (N=39)
Headache (Nervous system disorders) | 5 | 5 | 4 | 4 | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site vesicles (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.